CLINICAL TRIAL: NCT05739487
Title: Changes of Visual Field Defects After Selective Intra-arterial Thrombolysis for Central Retinal Artery Occlusion
Brief Title: Changes of Visual Field Defects After IAT for CRAO
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ping Fei, Associate professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2022-057-1
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Central Retinal Artery Occlusion; Visual Field; Intra-arterial Thrombolysis
MeSH Terms: conditions — Retinal Artery Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IAT therapy: patients with central retinal artery occlusion received selective intra-arterial thrombolysis
  Interventions: Procedure: selective intra-arterial thrombolysis

INTERVENTIONS:
Procedure: selective intra-arterial thrombolysis — IAT introduces rt-PA (50mg) directly into the ophthalmic circulation by super-selective microcatheterization

SUMMARY:
Central retinal artery occlusion (CRAO) is an ophthalmic emergency which leads to devastating visual function defects and poor prognosis. Though traditional conservative treatments are widely used, none of them is proved to be effective. A number of meta-analyses and observational studies indicate intravenous thrombolysis to be beneficial in CRAO. Selective intra-arterial thrombolysis (IAT) introducing rt-PA directly into the ophthalmic circulation by super-selective microcatheterization may reduce the complications such as intracranial and systemic hemorrhage. The residual visual field is significant for patients with CRAO who have poor central visual acuity. Thus, it is clinically significant to study the changes in visual fields in eyes with CRAO.

DETAILED DESCRIPTION:
Central retinal artery occlusion (CRAO) is an ophthalmic emergency which leads to devastating visual function defects and poor prognosis. Though traditional conservative treatments are widely used, none of them is proved to be effective. The respective responses of brain and retinal tissues to acute ischemia share many features is the rationale for therapeutic thrombolysis in CRAO. Intravenous thrombolysis (IVT) has been a therapeutic choice for CRAO since the 1960s, and in the United States, tPA is currently administered in 5.8% of patients admitted with CRAO. A number of meta-analyses and observational studies indicate intravenous thrombolysis to be beneficial in CRAO. Selective intra-arterial thrombolysis (IAT) introducing rt-PA directly into the ophthalmic circulation by super-selective microcatheterization which has the advantage of reducing the dose of rt-PA reaching the systemic circulation. It is clinically significant to study the changes in visual fields in eyes with CRAO. The short-term temporal changes (≤7-day) of VFDs and the adverse reactions in eyes with CRAO after IAT were investigated to assess the efficacy and safety of the procedure in this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Non-arteritic CRAO with symptom duration ≤7d 2. Age from 18 years old between 80 years old 3. Qualified systemic conditions, well-controlled blood pressure, well-controlled blood glucose, qualified liver and kidney function, no allergic history to contrast agent or rt-PA.

Exclusion Criteria:

* Ocular factor or disease

  1. Branch retinal artery occlusion
  2. Combined retinal vein occlusion
  3. Suspicious ocular ischemic syndrome, such as ophthalmic artery occlusion or carotid artery occlusion
  4. Existed retinal problems decreasing visual function, such as macular disease, severe nonproliferative or proliferative diabetic retinopathy, severe cataract or glaucoma
  5. Central retinal artery occlusion from iatrogenic cause
  6. History of thrombolysis for CRAO or CRVO
* Systemic factors restricting thrombolysis

  1. Uncontrolled hypertension (systolic blood pressure > 180mmHg ); Uncontrolled hyperglycemia (fasting blood glucose > 9mmol/L);
  2. Coagulation disorder
  3. History of intracranial hemorrhage, heart attack, cerebral infarction, or intracranial surgery within 3 mo
  4. Current antithrombotic treatment
  5. History of allergic reaction to contrast agent or rt-PA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-arteritic CRAO and treated by IAT between July 2020 and March 2022 were analyzed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change of the mean deviation | 7 days
  Change of the visual field index as mean deviation (MD) examed by Humphrey visual field analyzer at 7days
Change of the visual field index | 7 days
  Change of the visual field index as visual field index (VFI) examed by Humphrey visual field analyzer at 7 days

SECONDARY OUTCOMES:
Change of best corrected visual acuity (BCVA) | 7 days
  best corrected visual acuity of logarithm of the minimum angle of resolution
Adverse reactions at 7 days | 7 days
  Death, symptomatic or asymptomatic intracranial hemorrhage, intraocular hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Ping Fei, MD#PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided